CLINICAL TRIAL: NCT05527808
Title: Neoadjuvant Tislelizumab and Platinum-Based Doublet Chemotherapy in Stage II-IIIB EGFR-Mutated Lung Adenocarcinoma With PD-L1 Positive Expression -- A Phase II Study (DuoVitality)"
Brief Title: A Single-arm Exploratory Study of Neoadjuvant Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Liu (Other)
Responsible Party: Sponsor-Investigator, Jun Liu, Chief Physician, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tislelizumab-Neoadjuvant
Record Dates: First submitted 2022-08-03; First posted 2022-09-06 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Lung Adenocarcinoma
Keywords: Resectable II-IIIB; EGFR mutation and PD-L1≥1%; NSCLC; Neoadjuvant immunotherapy
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — tislelizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant ICI combined with chemotherory (Experimental): intravenous injection :Tislelizumab + pemetrexed + platinum Q3W 2-4 cycles
  Interventions: Drug: Tislelizumab; Drug: pemetrexed; Drug: cis-platemum; Drug: or carboplatin

INTERVENTIONS:
Drug: Tislelizumab — 200 mg ,intravenous injection ,Q3W 2-4 cycles
Drug: pemetrexed — 500 mg/m2,intravenous injection ,Q3W 2-4 cycles
Drug: cis-platemum — 60-75mg/m2 ,intravenous injection ,Q3W 2-4 cycles
Drug: or carboplatin — AUC(4-5) ,intravenous injection ,Q3W 2-4 cycles

SUMMARY:
Neoadjuvant EGFR TKI therapy targeting EGFR mutation has some problems failure to fulfill clinical requirements such as low MPR rate, tissue fibrosis and other major surgical impacts and unmet clinical needs.This study hypothesized that Tisleizumab combined with chemotherapy in the neoadjuvant treatment of stage II-IIIA non-squamous NSCLC with EGFR-mutant PD-L1 expression ≥1% could significantly improve the pathological response rate after neoadjuvant therapy, improve the surgical complete resection rate, reduce perioperative complications and do not increase the surgical difficulty.In this study, biomarker analysis is going to explore the possible direction of neoadjuvant therapy population screening, and to explore a possible method for the efficacy and safety of neoadjuvant immunotherapy in clinical stage II-IIIA non-squamous non-small cell lung cancer with EGFR mutation and expression of PD-L1.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research;Fully understand and be Informed of the study and sign the Informed Consent Form (ICF);Willing to follow and able to complete all test procedures;
2. Age 18-75 (boundary value included), no gender limitation;
3. Histologically proven stage II-IIIB Lung Adenocarcinoma (as defined by the American Joint Commission on Cancer, 8th Edition);
4. EGFR gene mutation positive (can be tested by tissue or blood samples);
5. PD-L1 ≥ 1%
6. ECOG PS score 0-1 (including boundary value);
7. Cardiopulmonary function is good, and the requirements for surgical resection for radical treatment are confirmed;
8. Meet the conditions for receiving platinum containing two-drug chemotherapy;
9. The expected survival time is ≥3 months, and feasible surgery is planned;

Exclusion Criteria:

1. Any previous treatment for current lung cancer, including systemic therapy or radiotherapy;
2. there are locally advanced unresectable diseases (regardless of disease stage) and metastatic diseases (stage IV).
3. A history of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc.Patients with any severe and/or uncontrolled disease or symptom

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response rate (MPR) （proportion of patients with no more than 10% remaining live tumor cells in the resected primary tumor and in all resected lymph nodes） | 15-18 weeks after enrollment
  MPR of surgical specimens from patients who were operable after neoadjuvant therapy was evaluated

SECONDARY OUTCOMES:
ORR: Proportion of patients who achieved complete response (CR) or partial response (PR) among all randomized patients with measurable disease at baseline assessed according to RECIST version 1.1 | 6-12weeks after enrollment
  To evaluate objective response rate (ORR) in neoadjuvant treatment
pCR: proportion of patients with no residual tumor in resected primary tumor and lymph nodes | 15-18 weeks after enrollment
  pCR of surgical specimens from patients who were operable after neoadjuvant therapy was evaluated
Descending rate of lymph nodes | 15-18 weeks after enrollment
  Proportion of patients whose pathologic lymph node stage was reduced to N1/N0 by baseline radiographic assessment of N2 or N1
Number of Participants with Adverse Events | through study completion, an average of 35weeks
  To evaluate the safety profile(Number of Participants with Adverse Events)
The time of surgery delay | 4-6weeks after completation of the last neoadjuvant therapy
  evaluate the interval time from the completation of last neoadjuvant therapy to surgery
minimally invasive surgery rate | 4-6weeks after completation of the last neoadjuvant therapy
  explore different surgery manner rate after neoadjuvant

CONTACTS AND LOCATIONS:
Overall Officials: Jun liu, Professor, Principal Investigator — 1First Affiliated Hospital, Guangzhou Medical University, Guangzhou, China
Locations (1):
- First Affiliated Hospital, Guangzhou Medical University, Guangzhou, Please Select, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chansky K, Detterbeck FC, Nicholson AG, Rusch VW, Vallieres E, Groome P, Kennedy C, Krasnik M, Peake M, Shemanski L, Bolejack V, Crowley JJ, Asamura H, Rami-Porta R; IASLC Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions. The IASLC Lung Cancer Staging Project: External Validation of the Revision of the TNM Stage Groupings in the Eighth Edition of the TNM Classification of Lung Cancer. J Thorac Oncol. 2017 Jul;12(7):1109-1121. doi: 10.1016/j.jtho.2017.04.011. Epub 2017 Apr 28. PMID 28461257
- [Background] Wozniak AJ, Gadgeel SM. Adjuvant therapy for resected non-small cell lung cancer. Ther Adv Med Oncol. 2009 Sep;1(2):109-18. doi: 10.1177/1758834009338634. PMID 21789116
- [Background] Rosell R, Lopez-Cabrerizo MP, Astudillo J. Preoperative chemotherapy for stage IIIA non-small cell lung cancer. Curr Opin Oncol. 1997 Mar;9(2):149-55. doi: 10.1097/00001622-199703000-00008. PMID 9161793
- [Background] Zhong WZ, Chen KN, Chen C, Gu CD, Wang J, Yang XN, Mao WM, Wang Q, Qiao GB, Cheng Y, Xu L, Wang CL, Chen MW, Kang X, Yan W, Yan HH, Liao RQ, Yang JJ, Zhang XC, Zhou Q, Wu YL. Erlotinib Versus Gemcitabine Plus Cisplatin as Neoadjuvant Treatment of Stage IIIA-N2 EGFR-Mutant Non-Small-Cell Lung Cancer (EMERGING-CTONG 1103): A Randomized Phase II Study. J Clin Oncol. 2019 Sep 1;37(25):2235-2245. doi: 10.1200/JCO.19.00075. Epub 2019 Jun 13. PMID 31194613
- [Background] NSCLC Meta-analysis Collaborative Group. Preoperative chemotherapy for non-small-cell lung cancer: a systematic review and meta-analysis of individual participant data. Lancet. 2014 May 3;383(9928):1561-71. doi: 10.1016/S0140-6736(13)62159-5. Epub 2014 Feb 25. PMID 24576776